CLINICAL TRIAL: NCT00506155
Title: A Phase II Clinical Trial of Neoadjuvant Chemotherapy With M-VAC Plus Avastin in Patients With Locally Advanced Urothelial Cancer
Brief Title: Neoadjuvant Chemotherapy With Methotrexate, Vinblastine, Adriamycin and Cisplatin (M-VAC) Plus Avastin in Patients With Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0620
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Results first posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Urothelial Cancer; Avastin; Bevacizumab; Cisplatin; Doxorubicin; Methotrexate; Vinblastine; M-VAC
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Bevacizumab; Cisplatin; Doxorubicin; Methotrexate; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant Chemotherapy with M-VAC + Avastin (Experimental): Avastin 10 mg/kg by vein over 90 minutes. Cisplatin 70 mg/m^2 by vein over 4 hours. Doxorubicin 30 mg/m^2 by vein over 15 minutes. Methotrexate 30 mg/m^2 by vein over 30 minutes. Vinblastine Sulfate 3 mg/m^2 by vein over 30 minutes.
  Interventions: Drug: Avastin; Drug: Cisplatin; Drug: Doxorubicin; Drug: Methotrexate; Drug: Vinblastine Sulfate

INTERVENTIONS:
Drug: Avastin — 10 mg/kg by vein over 90 minutes
  Other Names: Bevacizumab; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Cisplatin — 70 mg/m^2 by vein over 4 hours
  Other Names: Platinol-AQ; Platinol; CDDP
Drug: Doxorubicin — 30 mg/m^2 by vein over 15 minutes
  Other Names: Adriamycin; Rubex
Drug: Methotrexate — 30 mg/m^2 by vein over 30 minutes
Drug: Vinblastine Sulfate — 3 mg/m^2 by vein over 30 minutes

SUMMARY:
The goal of this clinical research study is to learn how well bladder cancer responds to a combination treatment with Avastin and M-VAC (methotrexate, doxorubicin, vinblastine, and cisplatin) before surgery to remove the tumor.

Primary Objective:

To estimate the response of patients with locally advanced urothelial cancer treated with neoadjuvant chemotherapy with a combination of Dose Dense Methotrexate, Vinblastine, Adriamycin, and Cisplatin (DD-M-VAC) plus Avastin followed by radical surgery with curative intent. In this context, response will be defined as the absence of residual muscle invasive cancer in the resected specimen (<= pT1, N0.)

Secondary Objective:

To estimate the 4-year disease-free survival of patients with locally advanced urothelial cancer treated with neoadjuvant chemotherapy with DD-M-VAC plus Avastin followed by radical surgery with curative intent.

Document perioperative morbidity and mortality in this cohort, with reference to well-established historical standards.

Determine the effects of VEGF inhibition on angiogenesis and angiogenesis-related gene expression utilizing fluorescent tissue staining techniques that we have developed in the laboratory (such as two-color TUNEL, phospho-receptor, and microvessel density).

Interrogate downstream receptor signaling pathways to provide insight into the development of chemotherapy resistance, and hence hypothesis for its prevention.

DETAILED DESCRIPTION:
Avastin is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels. Methotrexate, vinblastine, and doxorubicin are designed to disrupt the growth of cancer cells, which causes cancer cells to start to die. Cisplatin has an atom at its center that contains platinum. The platinum is designed to poison the cancer cells, which may cause them to eventually die.

If you are found to be eligible to take part in this study, you will be treated with the combination of Avastin, methotrexate, vinblastine, doxorubicin, and cisplatin. The study drugs and saline will be given through a needle in your vein. Avastin will be given over 90 minutes. Methotrexate will be given over 30 minutes. Vinblastine will be given over 30 minutes. Doxorubicin will be given over 15 minutes. Cisplatin will be given over 4 hours. You will also receive saline for hydration after you have completed the infusion of cisplatin. This will take up to 20 hours. If you have a catheter in place, the chemotherapy drugs as well as the saline will be given through the catheter. You will receive the study drugs 1 time every 2 weeks. Every 2 weeks is called a study "cycle".

On Day 1 of each cycle, you will have a physical exam, including measurement of your vital signs, height, and weight. You will be asked about any side effects you have experienced since your last visit. Blood (about 2 teaspoons) and urine will be collected for routine tests.

After 3 cycles of therapy, you will have a bone scan if your screening test showed signs of bone disease. You will also have a repeat cystoscopy. These tests will be done to check the status of the disease.

You will receive a total of 4 cycles of chemotherapy. At least 6 weeks after the last dose of Avastin, you will have a cystectomy (removal of your tumor). Your doctor will explain this procedure to you in detail. You will sign a separate consent form for this procedure.

After surgery, if you do not have disease in your lymph nodes or other sites, you will be taken off-study.

After surgery, if you still have disease in your lymph nodes or other sites, you will be eligible to continue treatment with Avastin. Therapy can be restarted no sooner than 28 days after your surgery. You will receive Avastin every 2 or 3 weeks through a needle in your vein. Every 2 or 3 weeks will be considered a study cycle.

Before each cycle of treatment, blood (about 1 teaspoon) will be drawn for routine tests. Urine will be collected every cycle for routine testing. Every 3 months you will have a CT scan or MRI to check the status of the disease.

You may continue to receive the study drug for up to 18 months of therapy. You will be taken off study in the disease gets worse or intolerable side effects occur.

Once you are off-study, you will have long term follow-up visits every 3-6 months for the first 30 months and then every year after that. These visits will continue for up to 4 years, or longer if your doctor thinks it is necessary. At these visits, you will have a CT or MRI scan of your abdomen and pelvis and a chest x-ray. Blood (about 1 teaspoons) will be drawn for routine testing.

This is an investigational study. Avastin is not FDA approved or commercially available for this indication. Its use in this study is considered to be investigational. Methotrexate, doxorubicin, vinblastine, and cisplatin are all FDA approved and commercially available. Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologic proof of urothelial cancer. Patients with all histologic subtypes are eligible as long as transitional cell carcinoma predominant, with 2 exceptions:

   * More than a few clusters of small cell carcinoma are treated with different chemotherapy and are ineligible for this study
   * Patients with micropapillary tumor will be allowed irrespective of the extent of transitional cell carcinoma. A transitional cell component is not required in the setting of pure or extensive micropapillary tumors. Note that minor histologic components are acceptable.
2. Patients with primary tumors arising in the bladder or urethra are eligible if they demonstrate any of the following features:

   * A 3-dimensional mass on examination under anesthesia (EUA); ie: cT3b disease
   * Direct invasion of prostatic stroma or the vaginal wall: ie:cT4a disease
   * Lymphovascular invasion on the specimen with >/= cT1 disease
   * Hydronephrosis present on CT scan or on renal ultrasound
   * Tumor involving bladder diverticulum.
3. Patients with more than a few areas of micropapillary histology are eligible, even if they do not meet the anatomic criteria for locally advanced disease enumerated above. Patients with micropapillary histology will be analyzed as a separate cohort.
4. Patients with primary tumors arising in the ureter or renal pelvis are eligible they have either grade 3 tumor, or a radiographic abnormality large enough to recognize as an abnormal mass by CT or MRI imaging. These patients may also be analyzed separately, since we do not have benchmark data for upper tract disease.
5. Patients must have an evaluation in the department of urology, and be deemed an acceptable surgical candidate.
6. Patients must have adequate physiologic reserves as by:

   * Zubrod performance status (PS) of </= 1; or 2 if of recent onset and due entirely to the cancer and not due to comorbidity (especially if the compromised performance status is related to uncontrolled pain which is expected to be rapidly reversible when therapy starts)
   * Normal WBC, ANC >/= 1,800, and platelet count >/= 150,000. Supranormal values judged to be of benign or inconsequential etiology are acceptable
   * Transaminase (AST or ALT) </= 3 * the ULN
   * Conjugated bilirubin </= 1.5 mg/dl (or total bilirubin </= 2.5 mg/dl)
   * Normal Serum Creatinine or Creatinine clearance (either measured or by Cockcroft-Gault formula) of >/= 50 ml/min.Cockcroft-Gault: CLcr = [(140-age) * wt(kg)]/[72 * Cr(mg/dL)] (For females, multiply by 0.85)
7. Patients (Pts) must NOT have clinical evidence of disease beyond the involved organ by either CT or MRI of the abdomen and pelvis, and chest X-ray. Pts with lymph node involvement are not eligible. In absence of a bone scan, pts should be free of bone pain and have an alk. phos. < 150% of the ULN, or a normal bone fraction of alk. phos. If these features are present, pts should have a bone scan and this should be interpreted as showing no evidence of metastatic disease to be eligible. In case of bladder tumors, cancer invading local organs (pT4a) but not pelvis sidewall (pT4b) are allowed.
8. Patients must have a determination of LV function with an EF >/= 50% to participate.
9. Women of child-bearing potential (i.e., who has had menses at any time in the preceding 24 consecutive months) must have a negative pregnancy test. Elevations of BHCG which are related to tumor (and not the rapid escalation associated with pregnancy, i.e. doubling time of 3-5 days) are acceptable.
10. Patients of child-bearing or child-fathering potential must agree to use an acceptable form of birth control while on the study, i.e. condoms.
11. Patients with second malignancies are eligible provided that the expected outcome from the second cancer is such that this will not interfere in the delivery of this therapy, or the assessment of response in the cystectomy specimen. The expected survival from the prior malignancy should reliably be > 4 years to be eligible for this study.
12. Patients must be >/= 18 years of age.

Exclusion Criteria:

1. Patients must not have current, recent (within 3 weeks), or planned participation with other experimental medication clinical trials.
2. Prior systemic cytoreductive chemotherapy for bladder cancer. Please note, that prior intra-vesical therapy is allowed.
3. Blood pressure of > 140/90 mmHg. Patients whose blood pressure is controlled with oral medication are eligible, as long as the blood pressure is </= 140/90 mmHg.
4. Any prior history of hypertensive crisis or hypertensive encephalopathy.
5. New York Heart Association (NYHA) Grade II or greater congestive heart failure.
6. History of myocardial infarction or unstable angina within 6 months prior to study enrollment.
7. History of stroke or transient ischemic attack within 6 months prior to study enrollment.
8. Clinically significant peripheral vascular disease (e.g., aortic aneurysm, aortic dissection).
9. Symptomatic peripheral vascular disease.
10. Evidence of bleeding diathesis or coagulopathy.
11. Known history of central nervous system or brain metastases.
12. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, anticipation of need for major surgical procedure during the course of the study. For the purpose of this study, Cystoscopy and ureteroscopy is not included as a major surgical procedure.
13. Lactating women.
14. Proteinuria at screening as demonstrated by either:

    * Urine protein:creatinine (UPC) ratio >/= 1.0 at screening OR
    * Urine dipstick for proteinuria > 2+ (or > 100 protein on urinalysis) Patients discovered to have >2+ proteinuria on dipstick urinalysis or >100 on urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate <= 1g of protein in 24 hours to be eligible.
15. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to therapy. Patients with Crohn's disease will be excluded.
16. Serious, non-healing wound, ulcer, or bone fracture.
17. Lung carcinoma of squamous cell histology or any histology in close proximity to a major vessel, cavitation, or history of hemoptysis (bright red blood of 1/2 teaspoon or more; non-small cell lung cancer trials only).
18. Inability to comply with study and/or follow-up procedures, or sign informed consent.
19. Patients who are not candidates for surgery, or are unwilling to undergo surgery.
20. Patients with fluid collections (such as ascites, or pleural effusions) are not eligible for therapy as such collections may serve as a reservoir for methotrexate.
21. Know hypersensitivity to any component of Avastin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Siefker-Radtke, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] McConkey DJ, Choi W, Shen Y, Lee IL, Porten S, Matin SF, Kamat AM, Corn P, Millikan RE, Dinney C, Czerniak B, Siefker-Radtke AO. A Prognostic Gene Expression Signature in the Molecular Classification of Chemotherapy-naive Urothelial Cancer is Predictive of Clinical Outcomes from Neoadjuvant Chemotherapy: A Phase 2 Trial of Dose-dense Methotrexate, Vinblastine, Doxorubicin, and Cisplatin with Bevacizumab in Urothelial Cancer. Eur Urol. 2016 May;69(5):855-62. doi: 10.1016/j.eururo.2015.08.034. Epub 2015 Sep 3. PMID 26343003
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 1, 2007 to December 13, 2010. All recruitment done at The University of Texas (UT) MD Anderson Cancer.
Groups:
- Neoadjuvant Chemotherapy With M-VAC + Avastin: Avastin 10 mg/kg intravenous (IV) over 90 minutes. Cisplatin 70 mg/m^2 IV over 4 hours. Doxorubicin 30 mg/m^2 IV over 15 minutes. Methotrexate 30 mg/m^2 IV over 30 minutes. Vinblastine Sulfate 3 mg/m^2 IV over 30 minutes.
Period: Overall Study
Arm/Group | Neoadjuvant Chemotherapy With M-VAC + Avastin
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Chemotherapy With M-VAC + Avastin
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 64 [42 to 79.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 60
Histology of Urothelial Cancer [Number; unit: participants] — Histological variants of urothelial tumors classified according to World Health Organization (WHO)/International Society of Urologic Pathologists (ISUP) 2004 guidelines; analysis by histologic types identified as TCC or divergent histologic differentiation (mixed histologic features).
  participants
    Transitional cell carcinoma (TCC) | 48
    Mixed | 12
    Mixed, Micropapillary | 8
Primary Site [Number; unit: participants] — Primary cancer site is location cancer starts in body. All participants with upper tract disease had high-grade disease and were N0M0. Since resection to the muscularis is not possible owing to the inherent risk of perforation in upper tract disease, cancer stage is not available in these participants.
  participants
    Renal Pelvis/Ureter | 16
    Bladder/Urethra | 44
Clinical Stage [Number; unit: participants] — Clinical cancer stage based on available information obtained before tumor removal surgery using "TNM"; T describes size of tumor and any spread of cancer into nearby tissue; N describes spread of cancer to nearby lymph nodes; & M describes metastasis (spread of cancer to other parts of body). Numbers after T (such as T1, T2, T3, and T4) describe tumor size and/or amount of spread into nearby structures, higher the T number, the larger the tumor and/or more it has grown into nearby tissues. All patients with T1 or T2 disease had high risk factor present to be eligible for trial.
  participants
    T1N0M0 | 4
    T2N0M0 | 13
    T3-4a N0M0 | 27
High risk feature [Number; unit: participants] — Low risk or high risk are based upon likelihood of cancer recurrence, including size, number, and appearance of tumor(s), if it recurs, and how deeply it invades into the bladder. A person whose cancer is low risk may be able to have less aggressive treatment and follow up, whereas a person with high risk bladder cancer may require more aggressive treatment and more frequent follow up. Participants may have more than one high-risk feature, so numbers exceed total number of participants.
  participants
    Lymphovascular invasion | 23
    Hydronephrosis | 20
    Diverticula | 1
    High-grade upper tract tumor | 16
    Three-dimensional mass on exam under anesthesia | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response Defined as the Absence of Residual Muscle Invasive Cancer in Resected Specimen
Description: Number of participants out of total with a response defined as "downstaging" to <= pT1N0 in the resected specimen. A binary variable was defined for downstaging (pathologic stage below initial clinical stage and below pT1N1N0M0); staging using American Joint Committee on Cancer (AJCC) TNM system of "TNM"; T describes size tumor & cancer spread into nearby tissue; N describes spread to nearby lymph nodes; & M describes metastasis (spread to other parts of body). Numbers after T (such as T1, T2, T3, and T4) describe tumor size and/or amount of spread into nearby structures, higher the T number, the larger the tumor and/or more it has grown into nearby tissues. Responses of lesser magnitude scored as treatment failure. Response Evaluation Criteria In Solid Tumors (RECIST) criteria do not apply for this cohort of neoadjuvant participants since this study does not require measurable disease by traditional assessment.
Time Frame: Following 20 weeks of chemotherapy
Population: All 60 participants completed at least 1 cycle of chemotherapy.
Measure: Number; unit: Percentage of Participants
Arm/Group | Neoadjuvant Chemotherapy With M-VAC + Avastin
Number analyzed (Participants) | 60
Percentage of Participants
  pT0N0 | 38
  pT1N0 | 53

2. Secondary Outcome: 5-year Overall Survival (OS)
Description: The overall survival rate stated as a five-year survival rate, which is the percentage of participants in study who are alive five years after the start of treatment.
Time Frame: 5 years
Measure: Number; unit: Percentage of Participants
Arm/Group | Neoadjuvant Chemotherapy With M-VAC + Avastin
Number analyzed (Participants) | 60
Percentage of Participants | 63

ADVERSE EVENTS:
Time Frame: Adverse event reporting collected through cystectomy performed at a minimum of 6 weeks from the last dose of Avastin.
Arm/Group | Neoadjuvant Chemotherapy With M-VAC + Avastin
Serious Adverse Events (participants affected / at risk) | 6/60
Other Adverse Events (participants affected / at risk) | 33/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Chemotherapy With M-VAC + Avastin (N=60)
Neutropenia/neutropenic fever (Infections and infestations) | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Chemotherapy With M-VAC + Avastin (N=60)
Neutropenia/neutropenic fever (Infections and infestations) | 10
Fatigue (General disorders) | 7
Hypertension (Cardiac disorders) | 4
Anemia (Blood and lymphatic system disorders) | 4
Thrombosis/pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Nausea/Vomiting (Gastrointestinal disorders) | 3
Mucositis (Gastrointestinal disorders) | 2
Thrombocytopenia (Skin and subcutaneous tissue disorders) | 2
Syncope (Nervous system disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Cardiac disorders) | 1
Transaminitis (Metabolism and nutrition disorders) | 1
Cardiac ischemia (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes